CLINICAL TRIAL: NCT02755584
Title: A Pilot Study of Skin Cells That Stop Replicating (Senescent) During Wound Healing
Brief Title: Study of Skin Cells That Stop Replicating (Senescent) During Wound Healing
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999916101; 16-AG-N101
Record Dates: First submitted 2016-04-28; First posted 2016-04-29 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2025-04-07

CONDITIONS: Healthy Volunteers
Keywords: Aging; Senescent Cells; Natural History

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: between the ages of 20-39 years and 70 years old and older

SUMMARY:
Background:

Cellular senescence is the aging of cells. It is a complex process that may be connected with aging and age-related diseases. It is unknown if these cells appear around wound sites in humans a few days after skin injury and if there are differences in young and old individuals. This study is being done to look at how cells in your body respond to small skin wounds. This information may help treat age-related diseases.

Objective:

To study how cells in the body respond to small skin wounds.

Eligibility:

Healthy adults ages 20-39 or 70+

Design:

Participants will be screened with medical history, physical exam, and blood sample. They will fast before the screening visit. Women will have a urine pregnancy test.

Participants will have 3 study visits over about 3 weeks.

Visits 1 and 2: Participants will fast before and have blood taken. Women will have a urine test. All participants will have 2 skin biopsies. A spot on the upper arm will be numbed. Two small pieces of skin will be removed. They will keep the area covered until the next visit.

Visit 3: Participants will have their vital signs taken. Their biopsy wounds will be measured and photographed.

DETAILED DESCRIPTION:
Objectives and Specific Aims:

The objective of this proof-of-concept study is to understand the physiological role of senescent cells in humans during the aging process using a model of wound healing. Cellular senescence is the phenomenon by which normal cells cease to divide in response to a stress. We aim to determine if in healthy humans: (1) senescent cells appear around wound sites a few days after skin injury; (2) the number of senescent cells induced by skin injury increases with age; (3) the wound healing process, as determined by the size of the healed wounds, is altered with aging; (4) biomarkers of senescence-associated secretory phenotype (SASP) increase significantly in the tissue around the wound a few days after skin injury, and the magnitude of increase is higher in older compared to younger persons; (5) ethnic differences in the dynamics of the appearance of senescent cells and whether such a difference is associated with wound healing. We also want to describe changes that occur with aging in DNA methylation and histone acetylation, gene expression, and protein expression within senescent cells in comparison to normal tissue.

Experimental Design and Methods:

One hundred and twenty-eight healthy participants, sixty-four between the ages of 20-39 years and sixty-four 70 years old or older will be recruited for this pilot study. Of the sixty-four participants in each age group, thirty-two will be men and thirty-two will be women and sixteen

will be Caucasian and sixteen will be African American. Each participant will have two 3mm skin biopsies on the inner upper arm during baseline visit (Visit 1) and two 6mm skin biopsies concentric to the previous site during Visit 2. Visit 2 will be scheduled on 8 different days (day 3, 5, 7, 9, 11, 13, 21 and 30) after the baseline visit with two men and two woman from each age/ethnic group for each of the days. A follow-up visit will be scheduled at the discretion of the medical staff. Senescent cells will be visualized by confocal microscopy based on a number of senescent markers described in the literature. Senescent biomarkers will be measured in the tissue and systemically at baseline and follow-up.

Medical Relevance and Expected Outcome:

Cellular senescence is a complex process characterized by arrest in replication that is thought to be intrinsically connected with aging and age-related diseases. Recently, researchers have

suggested that senescent cells may play a role in the pathogenesis of type 2 diabetes and its associated complications. Therefore, understanding the physiological role of senescent cells is critically important for understanding aging and age-related diseases such as type 2 diabetes. Preclinical data have shown that senescent cells were inducible during cutaneous wound healing. Our preliminary results showed that there may be a difference in rate of granulation tissue formation with ethnicity. Therefore, this method can be used to quantify

senescent cell response after a standard stimulus and to verify whether the magnitude of senescence response correlate with aging and ethnicity. In the future this method could be used to test interventions that can modify the senescence response, and may be an invaluable method for assessing novel treatments of type 2 diabetes involving senescent cells.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 20 - 39 years or age 70 years and older.
* Healthy (see exclusion criteria below).
* Are able to understand the study risks and procedures, and consent to participate in the study.
* Are able to read and speak English.
* Caucasian or African American
* Previous enrolled participants.

EXCLUSION CRITERIA (SCREENING VISIT):

* A medical condition that requires the use of chronic anticoagulant medication use such as warfarin, clopidogrel, heparin or antiplatelet agents other than low dose aspirin (81mg).
* History of increased bleeding due to either a known medical condition or an undiagnosed cause.
* A medical condition that causes impaired wound healing such as diabetes.
* Current androgenic/anabolic and/or corticosteroid use or use within 90 days of the procedure (ocular corticosteroid use okay).
* Current antibiotic or anti-viral use or use within 60 days of the procedure.
* Active infections or chronic skin conditions that would prevent access to the biopsy area.
* Taking non-steroidal anti-inflammatory agents (NSAIDs) such as Motrin (Ibuprofen), Advil (Ibuprofen) or Naprosyn (Naproxen) and the

participant is unable to stop taking them 3 days before the biopsy and 1 day after the biopsy procedure.

* Taking more than 81 mg of aspirin a day and the participant is unable to stop taking it for 3 days before the biopsy and 1 day after the biopsy procedure.
* Allergic to Lidocaine (Xylocaine) or any other local anesthetic or the participant has had in the past a severe allergic reaction to similar drugs.
* Allergic to topical betadine solution.
* Severe allergy to adhesives found in tape.
* HIV virus infection.
* Hepatitis B or C or exposure within 6 months of visit.
* History of diabetes (requiring any medical treatment other than diet and exercise) or fasting plasma glucose is >=126 mg/dL or HbA1c >= 6.5%.
* Clinically significant hormonal dysfunction (self-reported or laboratory values out of range. Mild hypothyroidism (TSH < 10 microIU/mL) in participants over 60 is not considered exclusion).
* Kidney disease (Creatinine >1.5 mg/dl or calculated creatinine clearance < 50 cc/min)
* Liver disease (Bilirubin > 1.5 mg/dl (unless higher levels can be ascribed to Gilbert s disease); ALT, AST or alkaline phosphatase twice the normal serum concentration).
* Severe gastrointestinal diseases such as Crohn s disease or ulcerative colitis requiring continuous treatment.
* History of severe pulmonary disease such as chronic obstructive pulmonary disease (COPD) or asthma requiring continuous medication use.
* History of severe psychiatric conditions associated with behavioral problems or requiring chronic medical treatment.
* Currently pregnant or breastfeeding.
* Participants with history of skin keloid formation during wound healing
* Current illness that as judged by the study physician substantially increases the risks associated the skin biopsy(s) (active infections, allergies, etc.).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes healthy volunteers between the ages of 20-39 years and 70 years old and older. Each age group will be men and women Caucasian and African American.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
To demonstrate that in humans, senescent cells will appear around wound sites after skin injury. | Basline visit 1and visit 2 six different days
  Understanding the physiological role of senescent cells is critically important for understanding aging and age related diseases. Our preliminary results showed that there may be a difference in rate of granulation tissue formation with ethnicity.

SECONDARY OUTCOMES:
The number of senescent cells induced by skin injury increases with age. The wound healing process, as determined by the size of the healed wounds, may be associated with aging. | ongoing
  The number of senescent cells induced by skin injury increases with age. The wound healing process, as determined by the size of the healed wounds, may be associated with aging.

CONTACTS AND LOCATIONS:
Overall Officials: Chee W Chia, M.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- National Institute on Aging, Clinical Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
The NIA IRP is discussing the plan to make IPD available. A final decision has not been made.